CLINICAL TRIAL: NCT04439071
Title: Evaluation of the Efficacy and Safety of PTC299 in Hospitalized Subjects With COVID-19 (FITE19)
Brief Title: A Study to Evaluate Efficacy and Safety of PTC299 (Emvododstat) in Hospitalized Participants With Coronavirus (COVID-19)
Acronym: FITE19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC299-VIR-015-COV19; 2020-001872-13 (EudraCT Number)
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Pneumonia; COVID-19; Coronavirus
MeSH Terms: conditions — Pneumonia; COVID-19; Coronavirus Infections | interventions — emvododstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTC299 + Standard of Care (SOC) (Experimental): Participants will receive PTC299 at 200 milligrams (mg), administered orally, twice daily (BID) on Days 1 to 7, then at 50 mg administered orally, once daily (QD) on Days 8 to 14.
  SOC will also be administered according to local, written policies or guidelines.
  Interventions: Drug: PTC299; Other: SOC
- Placebo + SOC (Placebo Comparator): Participants will receive PTC299-matching placebo administered orally, BID on Days 1 to 7, then administered orally, QD on Days 8 to 14.
  SOC will also be administered according to local, written policies or guidelines.
  Interventions: Other: SOC; Drug: Placebo

INTERVENTIONS:
Drug: PTC299 — Oral tablets
  Other Names: Emvododstat
  Arms: PTC299 + Standard of Care (SOC)
Other: SOC — As defined per local written policies or guidelines.
Drug: Placebo — Oral tablets
  Arms: Placebo + SOC

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter, 28-day study of adult participants hospitalized with COVID-19, with a safety follow-up telephone call at Day 60.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent document(s).
* Agrees to the collection of nasopharyngeal swabs and venous blood and all other protocol-specified procedures.
* Male or non-pregnant female adult ≥18 years of age at time of enrollment.
* Hospitalized and has laboratory-confirmed infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Symptom onset was ≤10 days prior to screening.
* Has oxygen saturation SpO2 <94% on room air.
* Has at least one of a respiratory rate >24 breaths/minute or cough.
* Lung involvement as confirmed by radiographic infiltrates observed on imaging (chest X-ray, computed tomography (CT) scan, or an equivalent test).
* Women of childbearing potential (as defined in [CTFG 2014]) must have a negative pregnancy test at screening and agree to abstinence or the use at least one of the following highly effective forms of contraception (with a failure rate of <1% per year when used consistently and correctly). Contraception or abstinence must be continued for the duration of the study following discharge from the hospital, and for up to 50 days after the last dose of study drug:

  i) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, and transdermal ii) progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, and implantable iii) intrauterine device iv) intrauterine hormone-releasing system v) vasectomized partner with confirmed azoospermia All females will be considered of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea in the appropriate age group without other known or suspected cause) or have been sterilized surgically (for example, bilateral tubal ligation, hysterectomy, bilateral oophorectomy).
* Men sexually active with women of childbearing potential who have not had a vasectomy must agree to use a barrier method of birth control during the study following discharge from the hospital and for up to 50 days after the last dose of study drug.

Exclusion Criteria:

* Requires mechanical ventilation.
* Current participation in any other interventional study.
* Alanine transaminase/aspartate transaminase levels ≥3 times the upper limit of normal (×ULN) or total bilirubin (Tbili) ≥2×ULN.
* Lymphocyte count <500 lymphocytes/microliter (μL) or hemoglobin <11 grams/deciliter (g/dL).
* Stage 4 severe chronic kidney disease or requiring dialysis (that is, estimated glomerular filtration rate <30).
* Any other condition, that in the opinion of the Investigator, may be cause to exclude the participant from the study.
* Use of steroids (except dexamethasone), sensitive CYP2D6 substrates, CYP2C inducers, IL-6 neutralizing antibodies, IL-6 receptor inhibitors, or any investigational therapy.
* Pregnancy or breast feeding.
* Anticipated transfer to another hospital which is not a study site within 72 hours.
* Known allergy to PTC299 or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quintus Ngumah, OD, PhD, Study Director — PTC Therapeutics
Locations (41):
- United States (6):
  - University of California, Irvine, Orange, California
  - Augusta University, Augusta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University Hospitals Cleveland, Cleveland, Ohio
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Hospital, St Albans, VC
  - Monash Medical Centre, Clayton, Victoria
- Belgium (2):
  - St. Pierre University Hospital, Brussels
  - Clinique Saint Pierre, Ottignies
- Brazil (8):
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Centro Hospitalar Unimed (CHU) - Joinville, Joinville, Santa Catarina
  - Hospital Guilherme Alvaro, Santos, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Escola Paulista de Medicina (UNIFESP), São Paulo, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São Paulo, São Paulo
  - Hospital Santa Casa de Misecórdia de Sorocoba, Sorocaba, São Paulo
- Colombia (2):
  - Fundación Santa Fe de Bogotá, Bogotá
  - Centro Cardiovascular Somer Incare, Rionegro
- Hôpital Pitié-Salpêtrière, Paris, France
- Mexico (4):
  - Centro Hospitalario MAC, Irapuato, Guanajuato
  - Hospital Universitario Dr. José Eleuterio Gonzalez, Monterrey, Nuevo León
  - Integra RGH Centro de Investigación/ Hospital MAC Puebla, Puebla City
  - SOMECO - Sociedad de Metabolismo y Corazón S.C., Veracruz
- Central Clinic Hospital of the MSWiA in Warsaw, Warsaw, Poland
- Portugal (3):
  - Centro Hospitalar Universitário de Lisboa Norte (CHULN), E.P.E - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de Entre o Douro e Vouga, EPE (CHEDV), Santa Maria da Feira
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE (CHVNG/E), Vila Nova de Gaia
- South Africa (5):
  - Worthwhile Clinical Trials, Benoni
  - TREAD Research, Cape Town
  - Tiervlei Trial Centre, Cape Town
  - Ahmed Al-Kadi Private Hospital, Durban
  - Global Clinical Trials, Pretoria
- Spain (6):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: FINAL REDACTED PROTOCOL — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217411&parentIdentifier=PTC299-VIR-015-COV19&attachmentIdentifier=642c87e2-eb4d-4a5c-85e5-1df1ccd361ef&fileName=Global_PTC299-VIR-015-COV19_Clinical_Protocol_V7.0_-_02JUN2021_final_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- PTC299: Participants received PTC299 at 200 milligrams (mg), administered orally, twice daily (BID) on Days 1 to 7, then at 50 mg administered orally, once daily (QD) on Days 8 to 14.
- Placebo: Participants received PTC299-matching placebo administered orally, BID on Days 1 to 7, then administered orally, QD on Days 8 to 14.
Period: Overall Study
Arm/Group | PTC299 | Placebo
Started | 94 | 95
Received at Least 1 Dose of Study Drug | 92 | 95
Completed | 80 | 77
Not Completed | 14 | 18
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Death | 6 | 4
Not completed — Other than specified | 3 | 3
Not completed — Randomized but not treated | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- PTC299: Participants received PTC299 at 200 mg, administered orally, BID on Days 1 to 7, then at 50 mg administered orally, QD on Days 8 to 14.
- Total: Total of all reporting groups
Arm/Group | PTC299 | Placebo | Total
Number analyzed (Participants) | 92 | 95 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (12.44) | 52.7 (12.48) | 52.3 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 67 | 68 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 64 | 117
  Not Hispanic or Latino | 34 | 26 | 60
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 1 | 7
  White | 69 | 69 | 138
  More than one race | 12 | 19 | 31
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Respiratory Improvement
Description: Respiratory improvement was defined as sustained peripheral oxygen saturation (SpO2) ≥94% on room air. Median time to respiratory improvement was estimated via the Kaplan-Meier product limit method.
Time Frame: up to Day 28
Population: Intent-to-treat (ITT) population included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 73 | 76
days | 10.0 [6.0 to 15.0] | 10.0 [8.0 to 13.0]
Statistical Analysis 1: Comparison: PTC299 vs Placebo; Time to respiratory improvement was compared between treatment groups using stratified log-rank test; Test type: Other; p = 0.949, Log Rank

2. Secondary Outcome: Number of Participants Requiring Invasive Ventilation
Description: Number of participants requiring invasive ventilation at any time during the study were reported.
Time Frame: up to Day 28
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 94 | 95
Participants | 16 | 11

3. Secondary Outcome: Number of Participants Requiring Supplemental Oxygen or Non-Invasive Ventilation in Participants Who Did Not Require Supplemental Oxygen at Baseline
Description: Number of participants requiring supplemental oxygen or non-invasive ventilation at any point during the study in participants who did not require supplemental oxygen at baseline were reported.
Time Frame: up to Day 28
Population: ITT population included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 24 | 22
Participants | 20 | 19

4. Secondary Outcome: Time From Randomization to Defervescence in Participants Presenting With Fever at Enrollment (Temperature of ≥37.6℃ Axilla, ≥38.0℃ Oral, or ≥38.6°C Tympanic or Rectal)
Description: Defervescence was defined as body temperature of <37.6° C axilla, <38.0° C oral, or <38.6° C tympanic or rectal without taking any antipyretic treatment and sustained until discharge or Day 28. Median time to defervescence was estimated via the Kaplan-Meier method.
Time Frame: up to Day 28
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 31 | 22
days | 7.0 [5.0 to 28.0] | 18.0 [4.0 to NA] — Due to smaller number of participants with an event, upper limit of 95% confidence interval (CI) could not be calculated.

5. Secondary Outcome: Time From Randomization to Respiratory Rate ≤ 24 Breaths Per Minute on Room Air
Description: Median time to respiratory rate in participants who had abnormal respiratory rate at baseline was estimated via the Kaplan-Meier method.
Time Frame: up to Day 28
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 57 | 62
days | 7.0 [5.0 to 11.0] | 8.0 [6.0 to 11.0]

6. Secondary Outcome: Time From Randomization to Cough Reported as Mild or Absent
Description: Cough was rated on a scale of severe, moderate, mild, absent, in those with cough at enrollment rated severe or moderate. Median time to cough reported as mild or absent was estimated via the Kaplan-Meier method.
Time Frame: up to Day 28
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 34 | 34
days | 3.0 [3.0 to 4.0] | 5.0 [3.0 to 7.0]

7. Secondary Outcome: Time From Randomization to Dyspnea Reported as Mild or Absent
Description: Dyspnea was rated on a scale of severe, moderate, mild, absent, in those with dyspnea at enrollment rated as severe or moderate. Median time to dyspnea reported as mild or absent was estimated via the Kaplan-Meier method.
Time Frame: up to Day 28
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 31 | 35
days | 6.0 [3.0 to 9.0] | 5.0 [4.0 to 7.0]

8. Secondary Outcome: Change From Baseline in Cytokine Levels at Day 28
Description: Cytokines included Granulocyte Colony Stimulating factor; Interleukin 10, 17, 2, 6, 7; Macrophage Inflammatory Protein 1 Alpha; Monocyte Chemotactic Protein 1; and Tumor Necrosis Factor.
Time Frame: Baseline, Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanograms (ng)/liter (L)
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 66 | 64
nanograms (ng)/liter (L)
  Granulocyte Colony Stimulating Factor | -0.423 (0.4431) | -0.467 (0.4750)
  Interleukin 10 | -0.367 (0.4655) | -0.491 (0.4003)
  Interleukin 17 | 0.018 (0.1447) | 0.002 (0.1425)
  Interleukin 2 | 0.021 (0.0868) | 0.022 (0.1448)
  Interleukin 6 | -0.375 (0.5274) | -0.442 (0.5062)
  Interleukin 7 | -0.025 (0.1233) | -0.035 (0.1556)
  Macrophage Inflammatory Protein 1 Alpha | 0.072 (0.2459) | 0.044 (0.1888)
  Monocyte Chemotactic Protein 1 | -0.011 (0.4077) | 0.018 (0.3804)
  Tumor Necrosis Factor | -0.015 (0.1509) | -0.027 (0.1666)

9. Secondary Outcome: Change From Baseline in Level of Acute Phase Protein (C Reactive Protein) at Day 28
Time Frame: Baseline, Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 51 | 46
mg/L | -1.027 (0.5966) | -1.111 (0.5633)

10. Secondary Outcome: Change From Baseline in Level of Acute Phase Protein (D-Dimer) at Day 28
Time Frame: Baseline, Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micrograms (µg)/L D-dimer units (DDU)
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 48 | 45
micrograms (µg)/L D-dimer units (DDU) | 0.029 (0.9278) | -0.121 (0.9392)

11. Secondary Outcome: Change From Baseline in Level of Acute Phase Protein (Ferritin) at Day 28
Time Frame: Baseline, Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: picomoles (pmol)/L
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 47 | 44
picomoles (pmol)/L | -0.410 (0.3096) | -0.497 (0.3162)

12. Secondary Outcome: Change From Baseline in Level of Acute Phase Proteins (Troponin I and Troponin T) at Day 28
Time Frame: Baseline, Day 28
Population: ITT population included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 32 | 18
µg/L
  Troponin I | 0.080 (1.5879) | -0.036 (0.2128)
  Troponin T: number analyzed (Participants) | 8 | 11
  Troponin T | 0.001 (0.0015) | 0.061 (0.1638)

13. Secondary Outcome: Number of Participants With Normalization of Complete Blood Count (CBC) Who Had CBC Out of Range at Baseline
Description: Number of participants who returned to normal range CBC were reported. CBC included red blood cell (RBC), hemoglobin (HGB), white blood cell (WBC), and Platelets.
Time Frame: up to Day 28
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 27 | 26
Participants
  RBC: number analyzed (Participants) | 13 | 18
  RBC | 7 | 13
  HGB: number analyzed (Participants) | 13 | 18
  HGB | 9 | 13
  WBC: number analyzed (Participants) | 27 | 19
  WBC | 22 | 17
  Platelets: number analyzed (Participants) | 26 | 26
  Platelets | 21 | 19

14. Secondary Outcome: Change From Baseline in Viral Load at Day 28: SARS-CoV-2 Immunoglobulin A (IgA) Antibody Ratio and SARS-CoV-2 Immunoglobulin G (IgG) Antibody Ratio
Time Frame: Baseline, Day 28
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 50 | 49
ratio
  SARS-CoV-2 IgA Antibody Ratio: number analyzed (Participants) | 49 | 49
  SARS-CoV-2 IgA Antibody Ratio | 0.003 (0.6387) | 0.165 (0.5122)
  SARS-CoV-2 IgG Antibody Ratio: number analyzed (Participants) | 50 | 47
  SARS-CoV-2 IgG Antibody Ratio | 0.890 (0.6846) | 0.874 (0.7604)

15. Secondary Outcome: Change From Baseline in Viral Load at Day 28: SARS-CoV-2 IgM Antibody Absorbance
Time Frame: Baseline, Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: absorbance (Abs)
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 45 | 47
absorbance (Abs) | 0.000 (0.4691) | 0.127 (0.4218)

16. Secondary Outcome: Change From Baseline in Viral Load at Day 28: SARS-CoV2 v2, SARS-CoV2 v2 Nasopharyngeal Swab (NPsw), and Severe Acute Resp Syndrome Coronavirus 2
Time Frame: Baseline, Day 28
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 4 | 2
copies/mL
  SARS-CoV2 v2: number analyzed (Participants) | 0 | 2
  SARS-CoV2 v2 |  | -0.345 (0.2235)
  SARS-CoV2 v2 NPsw: number analyzed (Participants) | 4 | 1
  SARS-CoV2 v2 NPsw | -1.201 (0.7503) | 1.532
  Severe Acute Resp Syndrome Coronavirus 2: number analyzed (Participants) | 1 | 0
  Severe Acute Resp Syndrome Coronavirus 2 | -0.432 |

17. Secondary Outcome: Duration of Hospitalization
Time Frame: up to Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 77 | 83
days | 8.1 (4.87) | 9.3 (5.49)

18. Secondary Outcome: Number of Mortalities at Day 28
Description: Mortality was defined as a death event occurring at anytime before the specific date, after the first dose has been received.
Time Frame: Day 28
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 92 | 95
Participants | 6 | 4

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. TEAEs were defined as any AEs that occurred on or after the first study treatment through 30 days after the last dose, or any AEs occurring before the first study treatment but worsening during the treatment through 30 days after the last dose. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: up to Day 60
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 92 | 95
Participants | 52 | 67

20. Other Pre Specified Outcome: Time From Randomization to Respiratory Improvement Where Symptom Onset Occurred ≤5 Days
Description: Respiratory improvement was defined as SpO2 ≥94% on room air. Median time to respiratory improvement was estimated via the Kaplan-Meier product limit method.
Time Frame: up to Day 28
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PTC299 | Placebo
Number analyzed (Participants) | 13 | 10
days | 10.0 [4.0 to 28.0] | 28.0 [7.0 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated.
Statistical Analysis 1: Comparison: PTC299 vs Placebo; Time to respiratory improvement was compared between treatment groups using stratified log-rank test; Test type: Other; p = 0.033, Log Rank

ADVERSE EVENTS:
Time Frame: up to Day 60
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | PTC299 | Placebo
All-Cause Mortality (participants affected / at risk) | 9/92 | 4/95
Serious Adverse Events (participants affected / at risk) | 21/92 | 24/95
Other Adverse Events (participants affected / at risk) | 50/92 | 63/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTC299 (N=92) | Placebo (N=95)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Septic shock (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 2 | 1
Pneumonia acinetobacter (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2
Disease progression (General disorders) | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PTC299 (N=92) | Placebo (N=95)
Alanine aminotransferase increased (Investigations) | 14 | 16
Aspartate aminotransferase increased (Investigations) | 12 | 12
Gamma-glutamyltransferase increased (Investigations) | 4 | 6
Constipation (Gastrointestinal disorders) | 10 | 12
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Anaemia (Blood and lymphatic system disorders) | 8 | 3
Lymphopenia (Blood and lymphatic system disorders) | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 2
Hypertension (Vascular disorders) | 7 | 2
Anxiety (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 2 | 6
Condition aggravated (General disorders) | 3 | 9
Headache (Nervous system disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04439071/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT04439071/SAP_001.pdf